CLINICAL TRIAL: NCT03267888
Title: Pilot Study of Pembrolizumab and Single-Fraction, Low-Dose, Radiation Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Pembrolizumab and Radiation Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097324; NCI-2017-01485 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4106-17 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: ISS Stage I Plasma Cell Myeloma; ISS Stage II Plasma Cell Myeloma; ISS Stage III Plasma Cell Myeloma; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation therapy, pembrolizumab (Experimental): Patients undergo radiation therapy on day 1. Patients also receive pembrolizumab IV over 30 minutes on day 2 or 3. Courses with pembrolizumab repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Pembrolizumab — Given 200 mg IV.
  Other Names: Keytruda; MK-3475
Radiation: Radiation Therapy — Patients will receive radiotherapy (8 Gy/1 fx) to an extra-osseous site and/or any bony site containing myeloma deposit.
  Other Names: Radiotherapy

SUMMARY:
This pilot clinical trial studies the side effects of pembrolizumab and radiation therapy in treating patients with stage I-III multiple myeloma that has come back after a period of improvement or that does not respond to treatment. Monoclonal antibodies, such as pembrolizumab, may block cancer growth in different ways by targeting certain cells. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving pembrolizumab and radiation therapy may work better in treating patients with stage I-III multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of concurrent single/low dose radiation therapy (radiotherapy) (8 Gy/1fx) in combination with pembrolizumab in relapsed or refractory myeloma patients.

SECONDARY OBJECTIVES:

I. To characterize late toxicity (Common Terminology Criteria for Adverse Events [CTCAE] > grade 2 toxicity at 6 and 12 months) and the effect of radiation in combination with pembrolizumab on systemic response rates using international myeloma working group (IMWG) uniform response criteria for multiple myeloma at 6 months and 12 months.

II. To assess changes in positron emission tomography/computed tomography (PET/CT) as a result of combining pembrolizumab and radiotherapy at 6 months and 12 months.

OUTLINE:

Patients undergo radiation therapy on day 1. Patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 2 or 3. Courses with pembrolizumab repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* International Staging System (ISS) stage I-III multiple myeloma that has progressive, relapsed, or refractory disease
* Able to give informed consent
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Relapsed and/or refractory myeloma; there is no minimum or maximum number of previous therapies that a patient may have received previously before being put on the current trial
* ≥ 1 osseous and/or extra-osseous lesion that can be radiated
* Candidate for pembrolizumab (as determined by physician, and adequate organ function)
* Candidate for radiotherapy (as determined by treatment physician); these patients can have symptomatic disease and/or asymptomatic disease; a minimum of one site of radiation is required to any osseous and/or any extra-osseous disease; radiation to any bony parts of the head and neck, skull, spine, ribs, and/or extremities are allowed; radiation to any bony part for documented lytic disease is allowed; radiation to any soft tissue plasmacytoma (including osseous and extra-osseous plasmacytoma) is allowed; the only exclusion criteria for radiation, is central nervous system (CNS) metastases
* Measurable myeloma disease (urine protein > 200 mg in 24 hours [hr] urine collection, serum free light chain ratio > 100 with an abnormal k/l ratio, serum M protein > 0.5 g/dl); 12 of the 24 patients do not have to have measurable disease
* Negative urine pregnancy test within 2 weeks for female subjects; female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
  * Abstinence is acceptable, if this is the usual life style and preferred contraception for the patient

Exclusion Criteria:

* Previous anti-programmed cell death protein 1 (PD1) or anti-PD-L1
* Solitary plasmacytoma
* Smoldering (asymptomatic) multiple myeloma
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency
* Known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its recipients
* Known additional malignancy that is progressing or requires active treatment (exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin)
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Known history of, or any evidence of active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; NOTE: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients requiring radiation for CNS diseases are excluded (CNS defined as brain soft tissue/intra parenchymal metastases within the gray and white matter of the brain and/or for cerebrospinal fluid [CSF] disseminated disease, including leptomeningeal carcinomatous disease)
* Has a history of allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K. Khan, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan MK, Nasti TH, Qian JY, Kleber TJ, Switchenko JM, Kaufman JL, Nooka AJ, Dhodapkar MV, Buchwald ZS, Obiekwe D, Lonial S, Ahmed R. Pembrolizumab and low-dose, single-fraction radiotherapy for patients with relapsed or refractory multiple myeloma: a prospective, single-centre, single-group, open-label, phase 2 pilot trial in the USA. Lancet Haematol. 2024 Jul;11(7):e510-e520. doi: 10.1016/S2352-3026(24)00105-4. Epub 2024 May 23. PMID 38797190
- See also: peer reviewed journal article — https://www-sciencedirect-com.proxy.library.emory.edu/science/article/pii/S2352302624001686?via%3Dihub

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy, Pembrolizumab: Patients undergo radiation therapy on day 1. Patients also receive pembrolizumab IV over 30 minutes on day 2 or 3. Courses with pembrolizumab repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Pembrolizumab: Given 200 mg/kg IV.
  Radiation Therapy: Patients will receive radiotherapy (8 Gy/1 fx) to an extra-osseous site and/or any bony site containing myeloma deposit.
Period: Overall Study
Arm/Group | Radiation Therapy, Pembrolizumab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy, Pembrolizumab
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 62 [48 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Greater than grade 2 toxicity will be assessed by Common Terminology Criteria for Adverse Events.
Time Frame: Up to 12 months after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy, Pembrolizumab
Number analyzed (Participants) | 25
Participants | 8

2. Secondary Outcome: Number of Patients Achieving Any Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR according to International Myeloma Working Group (IMWG) criteria.
Time Frame: Up to 12 months after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy, Pembrolizumab
Number analyzed (Participants) | 25
Participants | 8

3. Secondary Outcome: Number of Participants Who Showed an Overall Response to Treatment Based on Baseline Changes on Positron Emission to Positron Emission Tomography/Computed Tomography
Description: Will be defined using International IMWG criteria.
Time Frame: Up to 12 months after study start
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Radiation Therapy, Pembrolizumab
Number analyzed (Participants) | 25
participants | 20 [7 to 41]

4. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier product-limit method.
Time Frame: From first treatment on course 1, day 1 to the earlier of date of death and/or last follow up, assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Radiation Therapy, Pembrolizumab
Number analyzed (Participants) | 25
participants | 15

ADVERSE EVENTS:
Time Frame: The first 12 months of treatment
Arm/Group | Radiation Therapy, Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 10/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy, Pembrolizumab (N=25)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy, Pembrolizumab (N=25)
Fatigue (General disorders) | 4 (4)
Fever (Immune system disorders) | 2 (2)
Rigours during infusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03267888/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03267888/ICF_000.pdf